CLINICAL TRIAL: NCT02306018
Title: Evaluation of a New Calibrated Pulse Wave Analysis Method(EV1000™/volumeView™) for Cardiac Output Monitoring in Adult Liver Transplantation
Brief Title: Evaluation of EV1000™/volumeView™ for Cardiac Output Monitoring in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gwak Mi Sook, professor, Samsung Medical Center
Other Study IDs: 2014-08-080-002
Record Dates: First submitted 2014-10-17; First posted 2014-12-03 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Liver Disease
Keywords: liver transplantation; cardiac output
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EV1000™/volumeView™
  Interventions: Device: EV1000™/volumeView™

INTERVENTIONS:
Device: EV1000™/volumeView™

SUMMARY:
The investigators are trying to evaluate the agreement of cardiac output measurements taken using the specific thermistor-tipped arterial catheter ( the VolumeView ™ catheter) and the EV1000 ™ monitoring platform ( Edward lifesciences, Irvine, CA, USA) with measurements taken using continuous pulmonary artery thermodilution cardiac output monitoring during orthotopic liver transplantation.

DETAILED DESCRIPTION:
In cirrhotic patient undergoing liver transplantation, there are an altered patterm of circulation, which is characterized by increased cardiac output, decreased peripheral vascular resistance, and reduced ventricular response to physiological, pharmacological, and surgical stress. Large blood loss and clamping/declamping of the inferior vena cava and portal vein during liver transplantation surgery can affect intravascular volume status, which in turn can lead to hemodynamic instability. Therefore, reliable cardiac output monitoring is particularly useful in the cirrhotic patient undergoing liver transplant. Pulmonary artery thermodilution has been used as a standard method for cardiac output assessment for many years. Pulmonary artery catheter can cause rare but serious complications. And it has some limitations for continuously monitoring cardiac output during rapid hemodynamic changes.

Recently, several minimally invasive CO monitors have been developed. The pulse contour technique continuously estimates CO through mathematical analysis of the waveform of arterial pressure. However, previous studies evaluating the reliability of the pulse contour techniques indicated conflicting results in cirrhotic patients during liver transplantation. Most of studies were performed by analyzing from radial artery pressure waveform. Because of rapid changing of intravascular volume, using inotropics, the monitoring of femoral artery pressure has been recommended during liver transplantation.

A new pulse wave analysis system has developed and introduced into clinical practice that consists of a specific thermistor -tipped femoral arterial catheter ( the VolumeView™ catheter) and the EV1000™ monitoring platform ( Edward lifesciences, Irvine, CA, USA). To continuously assess CO based on the femoral arterial pressure curve signal and it uses transpulmonary thermodilution for calibration. We are trying to evaluate the agreement of cardiac output measurements taken using EV1000™ / VolumeView™ with measurements taken using continuous pulmonary artery thermodilution cardiac output monitoring during orthotopic liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

subjects undergoing living donor liver transplantation during the study period subjects older than 20yrs who can give informed consent

Exclusion Criteria:

those who are confirmed moderate severe aortic regurgitation by echocardiography those with infection on cannulation site

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are performed liver transplantation in Samsung medical center
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
cardiac output | intraoperative
  L/minute, 28 participants, EV1000 by femoral artery, Pulmonary artery thermodilution

SECONDARY OUTCOMES:
systemic vascular resistance | intraoperative
  dyne s/cm5,28 participants, EV1000 by femoral artery, Pulmonary artery thermodilution
stroke volume variability | during surgery every 10 minute, event time for example, anhepatic, liver in, reperfusion, using inotropics, changing ventilator setting
  %, 28 participants, EV1000 by femoral artery, Pulmonary artery thermodilution
stroke volume | intraoperative
  ml, 28 participants, EV1000 by femiral artery, Pulmonary artery thermodilution
ejection fraction | intraoperative
  %, 28 participants, EV1000 by femoral artery, Pulmonary artery thermodilution

CONTACTS AND LOCATIONS:
Overall Officials: Mi Hye Park, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Feltracco P, Biancofiore G, Ori C, Saner FH, Della Rocca G. Limits and pitfalls of haemodynamic monitoring systems in liver transplantation surgery. Minerva Anestesiol. 2012 Dec;78(12):1372-84. Epub 2012 Aug 3. PMID 22858882
- [Result] Uemura K, Kawada T, Inagaki M, Sugimachi M. A minimally invasive monitoring system of cardiac output using aortic flow velocity and peripheral arterial pressure profile. Anesth Analg. 2013 May;116(5):1006-1017. doi: 10.1213/ANE.0b013e31828a75bd. Epub 2013 Mar 14. PMID 23492964
- [Result] Biancofiore G, Critchley LA, Lee A, Bindi L, Bisa M, Esposito M, Meacci L, Mozzo R, DeSimone P, Urbani L, Filipponi F. Evaluation of an uncalibrated arterial pulse contour cardiac output monitoring system in cirrhotic patients undergoing liver surgery. Br J Anaesth. 2009 Jan;102(1):47-54. doi: 10.1093/bja/aen343. PMID 19059920
- [Result] Biancofiore G, Critchley LA, Lee A, Yang XX, Bindi LM, Esposito M, Bisa M, Meacci L, Mozzo R, Filipponi F. Evaluation of a new software version of the FloTrac/Vigileo (version 3.02) and a comparison with previous data in cirrhotic patients undergoing liver transplant surgery. Anesth Analg. 2011 Sep;113(3):515-22. doi: 10.1213/ANE.0b013e31822401b2. Epub 2011 Jun 16. PMID 21680855
- [Result] Tsai YF, Su BC, Lin CC, Liu FC, Lee WC, Yu HP. Cardiac output derived from arterial pressure waveform analysis: validation of the third-generation software in patients undergoing orthotopic liver transplantation. Transplant Proc. 2012 Mar;44(2):433-7. doi: 10.1016/j.transproceed.2011.12.045. PMID 22410036
- [Result] Galluccio ST, Chapman MJ, Finnis ME. Femoral-radial arterial pressure gradients in critically ill patients. Crit Care Resusc. 2009 Mar;11(1):34-8. PMID 19281442
- [Result] Arnal D, Garutti I, Perez-Pena J, Olmedilla L, Tzenkov IG. Radial to femoral arterial blood pressure differences during liver transplantation. Anaesthesia. 2005 Aug;60(8):766-71. doi: 10.1111/j.1365-2044.2005.04257.x. PMID 16029225
- [Result] Kim YK, Shin WJ, Song JG, Jun IG, Kim HY, Seong SH, Hwang GS. Comparison of stroke volume variations derived from radial and femoral arterial pressure waveforms during liver transplantation. Transplant Proc. 2009 Dec;41(10):4220-8. doi: 10.1016/j.transproceed.2009.09.050. PMID 20005373
- [Result] Sakka SG, Kozieras J, Thuemer O, van Hout N. Measurement of cardiac output: a comparison between transpulmonary thermodilution and uncalibrated pulse contour analysis. Br J Anaesth. 2007 Sep;99(3):337-42. doi: 10.1093/bja/aem177. Epub 2007 Jul 4. PMID 17611251
- [Result] Bendjelid K, Marx G, Kiefer N, Simon TP, Geisen M, Hoeft A, Siegenthaler N, Hofer CK. Performance of a new pulse contour method for continuous cardiac output monitoring: validation in critically ill patients. Br J Anaesth. 2013 Oct;111(4):573-9. doi: 10.1093/bja/aet116. Epub 2013 Apr 26. PMID 23625132
- [Result] Kiefer N, Hofer CK, Marx G, Geisen M, Giraud R, Siegenthaler N, Hoeft A, Bendjelid K, Rex S. Clinical validation of a new thermodilution system for the assessment of cardiac output and volumetric parameters. Crit Care. 2012 May 30;16(3):R98. doi: 10.1186/cc11366. PMID 22647561
- [Result] Bendjelid K, Giraud R, Siegenthaler N, Michard F. Validation of a new transpulmonary thermodilution system to assess global end-diastolic volume and extravascular lung water. Crit Care. 2010;14(6):R209. doi: 10.1186/cc9332. Epub 2010 Nov 23. PMID 21092252